CLINICAL TRIAL: NCT02744287
Title: A Phase 1/2 Feasibility, Safety, and Activity Study of PSCA-Specific Chimeric Antigen Receptor Engineered T Cells (BPX-601) in Subjects With Previously Treated Advanced Solid Tumors
Brief Title: Safety and Activity Study of PSCA-Targeted CAR-T Cells (BPX-601) in Subjects With Selected Advanced Solid Tumors
Status: Suspended | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Due to a Dose Limiting Toxicity.
Sponsor: Bellicum Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BP-012
Record Dates: First submitted 2016-04-11; First posted 2016-04-20 (Estimated); Last update posted 2023-04-20 (Actual); Status verified 2023-04

CONDITIONS: Metastatic Castration-resistant Prostate Cancer; Metastatic Prostate Cancer
Keywords: prostate stem cell antigen; BPX-601; AP1903; CAR-T; PSCA-CAR; castration-resistant prostate cancer; rimiducid; prostate cancer; PSCA; CRPC; mCRPC
MeSH Terms: conditions — Prostatic Neoplasms | interventions — AP 1903 reagent

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1: Phase 1 Dose Escalation (Experimental): Participants with advanced prostate cancer will receive an intravenous infusion of BPX-601 followed by one or more intravenous infusions of rimiducid. Dose escalation of BPX-601 will continue until the recommended cell dose level is reached.
  Interventions: Biological: BPX-601; Drug: Rimiducid
- Arm 2: Phase 2 Dose Expansion (Experimental): Participants with advanced prostate cancer will receive an intravenous infusion of BPX-601 at the recommended cell dose level followed by one or more intravenous infusions of rimiducid.
  Interventions: Biological: BPX-601; Drug: Rimiducid

INTERVENTIONS:
Biological: BPX-601 — Autologous T cells genetically modified with retrovirus vector containing PSCA-specific CAR and an inducible MyD88/Cluster Designation (CD)40 (iMC) co-stimulatory domain
Drug: Rimiducid — Dimerizer infusion to activate the iMC of the BPX-601 cells for improved proliferation and persistence
  Other Names: AP1903

SUMMARY:
The purpose of this study is to evaluate the safety and activity of BPX-601 CAR-T cells in participants with previously treated advanced solid tumors (prostate) expressing high levels of prostate stem cell antigen (PSCA). Participants' T cells are modified to recognize and target the PSCA tumor marker on cancer cells.

DETAILED DESCRIPTION:
The goal of this study is to characterize the feasibility, safety, and clinical activity of PSCA-specific CAR-T cells, BPX-601, administered with rimiducid to subjects with previously treated, PSCA-positive advanced solid tumors (prostate). BPX-601 CAR-T cells are genetically engineered to express a chimeric antigen receptor (CAR) to target the PSCA antigen and a rimiducid-inducible signaling domain which functions as a molecular "go-switch" to enhance activation and proliferation.

Phase 1: Cell dose escalation to identify the maximum dose of BPX-601 administered with single or repeat doses of rimiducid.

Phase 2: Indication-specific dose expansion to assess the safety, pharmacodynamics (including BPX-601 persistence), and clinical activity at the recommended dose identified in Phase 1 in various PSCA-expressing solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic castration-resistant prostate cancer (mCRPC), with progressive disease per PCWG3 criteria during or following the direct prior line of therapy.
* Measurable disease per RECIST v1.1 at baseline; subjects with mCRPC with bone only metastases must have measurable PSA.
* Age ≥18 years.
* Life expectancy > 12 weeks.
* ECOG 0-1
* Adequate organ function.

Exclusion Criteria:

* Prostate cancer with unstable bone lesions or symptomatic/untreated coagulopathy, or history of > Grade 2 hematuria within the previous 6 months.
* Prior CAR T cell or other genetically-modified T cell therapy. Prior treatment with an immune-based therapy for the treatment of prostate cancer, including cancer vaccine therapies are allowable.
* Symptomatic, untreated, or actively progressing central nervous system metastases.
* Impaired cardiac function or clinically significant cardiac disease.
* Pregnant or breastfeeding.
* Participant requires chronic, systemic steroid therapy.
* Severe intercurrent infection.
* Known HIV positivity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Estimated)
Dates: Start 2016-11 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicity | 4 weeks after first rimiducid infusion (i.e., Day 35)
  Incidence of dose limiting toxicity
Treatment emergent adverse events (AEs) and serious AEs (SAEs) | 180 days after BPX-601 treatment up to 15 years
  Number of participants with adverse events (AEs) and serious AEs (SAEs) assessed for severity using NCI CTCAE v4.03
Maximum tolerated dose (MTD) and/or recommended phase 2 dose (RP2D) | through Phase 1 completion, up to 5 years
  Identify the optimal dose of BPX-601 with rimiducid for Phase 2

SECONDARY OUTCOMES:
Pharmacodynamics (PD) of BPX-601 | up to 1 year after treatment
  Change from baseline in pharmacodynamic blood biomarkers - markers of BPX-601 CAR-T cells
Antitumor activity of BPX-601 | From the time of BPX-601 cell infusion until confirmed disease progression or death due to any cause, the start of new anticancer therapy, or withdrawal, whichever comes first, as assessed for up to 5 years after the last subject has been enrolled
  Percentage of subjects with objective response determined by the investigator according to the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 or the Prostate Cancer Working Group 3 (PCWG3) criteria

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - Moffitt Cancer Center, Tampa, Florida
  - Emory Winship Cancer Institute, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - University of Chicago Medicine, Chicago, Illinois
  - Karmanos Cancer Institute, Detroit, Michigan
  - University of Nebraska, Omaha, Nebraska
  - John Theurer Cancer Center, Hackensack University Medical Center, Hackensack, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Columbia University Medical Center, New York, New York
  - Duke University, Durham, North Carolina
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Baylor Sammons Cancer Center, Dallas, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stein MN, Dumbrava EE, Teply BA, Gergis US, Guiterrez ME, Reshef R, Subudhi SK, Jacquemont CF, Senesac JH, Bayle JH, Scripture CD, Chatwal MS, Bilen MA, Stadler WM, Becerra CR. PSCA-targeted BPX-601 CAR T cells with pharmacological activation by rimiducid in metastatic pancreatic and prostate cancer: a phase 1 dose escalation trial. Nat Commun. 2024 Dec 30;15(1):10743. doi: 10.1038/s41467-024-53220-6. PMID 39737899